CLINICAL TRIAL: NCT01992068
Title: Prospective Pilot Study of High-resolution Manometry to Assess Radiation-induced Changes in Esophageal Function in Patients With Lung Cancer
Brief Title: Pilot Study: Utilizing Manometry to Assess Radiation-Induced Changes in Esophageal Function
Status: Terminated | Type: Observational
Why Stopped: Closure due to low accrual
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: LCCC 1309; LCCC 1309 (Other Grant/Funding Number: Lineberger Comprehensive Cancer Center); 13-1113 (Other: UNC IRB)
Record Dates: First submitted 2013-11-18; First posted 2013-11-25 (Estimated); Last update posted 2017-04-06 (Actual); Status verified 2017-04

CONDITIONS: Lung Cancer
Keywords: lung cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Lung cancer patients ≥ 18 years of age: Lung cancer patients age ≥ 18 years or older who have:
  * Histologically confirmed lung cancer scheduled to undergo conventionally fractionated radiation treatment
  * Absence of any severe disorders of esophageal motility (patients with reflux and/or a hiatal hernia are eligible)

SUMMARY:
The purpose of this study is to prospectively assess the feasibility of high-resolution manometry to identify radiation-induced changes in esophageal motility and contractility or "function" in patients undergoing radiation therapy for the treatment of locally advanced lung cancer.

DETAILED DESCRIPTION:
As there is no standard of care to evaluate/visualize the effects of radiation therapy (RT) -induced esophageal injury, this is routinely assessed by patient reported accounts, and the symptoms are then managed supportively (e.g. with pain medicines, parenteral nutrition, feeding tubes etc). Manometry has been frequently used to study the effects of RT on gastrointestinal function in the setting of numerous malignancies, including colorectal, cervical and prostate cancers. What is often seen after RT is decreased sphincter function in the anorectal region leading to problems with continence and fecal urgency, however there has not been as rigorous of an evaluation of esophageal function after RT.

One study performed more than 15 years ago included only 4 patients with lung cancer and concluded that mucosal irritation was likely the primary cause of RT-associated esophageal injury and no abnormalities in motility were seen. Radiation is known to cause long-term esophageal injury including stricture, and there is manometric evidence of impaired motility long-term after RT. The recent introduction of high-resolution manometry permits more extensive evaluation of the effects of RT on esophageal function.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years or older
* Absence of any severe disorders of esophageal motility (patients with reflux and/or a hiatal hernia are eligible)
* Histologically confirmed lung cancer scheduled to undergo conventionally fractionated radiation treatment
* Patients that will be treated with a minimum of 45 Gy of radiation therapy
* Patients with mediastinal nodal disease, or primary lesions that are near the esophagus are eligible provided that they are not having esophageal symptoms believed to be due to the tumor.

Exclusion Criteria:

* History of esophageal motility disorder that pre-dates and is unrelated to the present diagnosis of lung cancer
* History of any prior radiotherapy to the esophagus
* Pregnant or lactating women
* Inability to understand and follow swallowing instructions for the esophageal manometry procedure; this is to ensure patient compliance of performing the breath hold technique throughout the radiation therapy treatment
* Patients with mediastinal nodal disease, or primary lesions, that are having esophageal symptoms believed to be due to the tumor

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lung cancer patients age 18 or above who have a histologically confirmed lung cancer diagnosis and are scheduled to undergo conventionally fractionated radiation treatment.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2013-09; Primary Completion 2016-12-12 (Actual); Study Completion 2016-12-12 (Actual)

PRIMARY OUTCOMES:
Utilizing manometry to assess radiation-induced changes to esophageal function | 6 months
  To evaluate the feasibility of high-resolution manometry to identify radiation-induced changes in esophageal function in patients undergoing radiation therapy for the treatment of locally advanced lung cancer.

SECONDARY OUTCOMES:
Rate of radiation-induced changes in esophageal function | 6 months
  To estimate the rate of radiation-induced changes in regional esophageal function.

OTHER OUTCOMES:
Associated changes in esophageal function: manometry versus the Mayo Dysphagia questionnaire | 6 months
  To explore the association of the changes in regional esophageal function during and after RT with changes in esophageal symptoms as assessed by the Mayo Dysphagia Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Zagar, MD, Principal Investigator — Department of Radiation Oncology, University of North Carolina Chapel Hill; Ryan Madanick, MD, Principal Investigator — Department of Medicine, University of North Carolina Chapel Hill
Locations (1):
- Department of Radiation Oncology Clinic, Chapel Hill, North Carolina, United States